CLINICAL TRIAL: NCT02044770
Title: Initial Clinical Experience With the ENSEAL® G2 Articulating Tissue Sealer in Laparoscopic Colectomy
Brief Title: ENSEAL® G2 Articulating Tissue Sealer in Laparoscopic Colectomy
Status: Completed | Type: Observational
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Other Study IDs: ENG 13-001
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2014-09

CONDITIONS: Any Condition Requiring Surgical Treatment Via Colectomy
Keywords: laparoscopic; colectomy; ENSEAL

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this clinical study is to describe the initial clinical experience with ENSEAL® G2 Articulating Tissue Sealer in laparoscopic colectomy, quantifying and/or qualifying how its articulation feature enables optimization of vessel sealing through improved access, approach, and visibility. This is an observational study of device usage being conducted to report initial experience with the ENSEAL ART device. It is not intended as hypothesis testing.

DETAILED DESCRIPTION:
The ENSEAL® G2 Tissue Sealer is a sterile, single-patient use surgical instrument used to coagulate and transect vessels up to and including 7mm in diameter and tissue and/or vascular bundles. In preclinical research using ENSEAL tissue sealers, burst pressures were 51% higher for perpendicularly sealed vessels than for angled seals (p<0.001) and the seal length was the primary variable in determining burst pressure (Voegele AC, 2013). These results suggest that the strongest possible seal may be obtained when vessels are approached perpendicularly and not at an angle.

However, desired angles for vessel sealing cannot always be obtained in the surgical field, especially in laparoscopic surgery due mostly to the fixed nature of the abdominal wall cannulas and the lack of adequate articulating hemostatic tools.

Since strong vessel seals are important for adequate homeostasis, the value of an articulating vessel-sealing device primarily resides in its ability to maneuver around corners and behind structures in confined spaces. An articulating vessel-sealing device would maximize the ability to approach vessels or bundles in a perpendicular manner to provide greater seal strength.

ENSEAL ART is the first articulating advanced bipolar device that can facilitate laparoscopic surgery through a 5mm port. The instrument shaft, can achieve up to 110 degrees of articulation (which improves the visibility of the tip of the device's jaw) to gain access to tissue in challenging anatomy, especially in deep/tight spaces, and facilitate additional angles to transect and seal tissue, vessels, and vascular bundles.

The articulation feature and improved ergonomics of the ENSEAL ART may provide the ability to maneuver around corners and behind structures, while making it easier to capture the full vessel in a single bite. These features may lead to a reduction of the number of ports, the instrument exchanges between ports, the need to pass the energy device to an assistant, and the number of times the surgical table tilt has to be changed during certain laparoscopic surgical procedures (e.g., colectomy).

This study focuses primarily in reporting initial user-centered interactions with the ENSEAL ART device. The users of the device will be board-certified colorectal surgeons, who will use it in an actual clinical setting (i.e., laparoscopic colectomies).

After obtaining Institutional Review Board approval, the study sites will begin recruitment of study participants.

At each of the participating study sites, 8 to 14 participants will undergo a laparoscopic colectomy using the ENSEAL ART for vessel dissection and sealing, according to the institution's standard approach.

Video recordings from the laparoscope and external cameras will capture all device activations completed with the ENSEAL ART device using articulation vs. straight (without articulating). After each surgical case, PIs will complete a survey related to the perceived advantages of the articulating features of ENSEAL ART in the context of their experience using non-articulation tissue sealers. PIs will also complete an assessment (using a validated tool) of the perceived workload of the use of the ENSEAL ART device.

The digital video recording of the surgical procedure will be evaluated by a consultancy group - Design Science Consulting Inc. (Philadelphia, PA), specializing in the conduct of field research of the variables pre-established by the protocol. Design Science is a third party reviewer, not associated with any of the study sites.

Subject-related data to be collected is limited to age, gender, diagnosis, Medical History, and adverse events associated to the use of the device.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (age ≥ 18 and < 80 years of age, on the day of the procedure
* Scheduled to undergo one of the following planned colectomies, anticipated to be performed laparoscopically:

  a. Right colectomy; b. Left hemicolectomy; c. Transverse colectomy; d. Sigmoidectomy; e. Total colectomy; or f. Subtotal colectomy. f. Subtotal colectomy.

Exclusion Criteria:

* Unable or unwilling to sign the study informed consent form;
* Previous colectomy and/or proctectomy;
* Anticipated combinations of laparoscopic colectomy and low anterior resection, except in cases in which the lower anterior resection is intended to be done with an energy device other than the ENSEAL® G2 Articulating Tissue Sealer;
* Any previous major surgery of the colon that, in the opinion of the surgeon, may increase the risk of intraoperative conversion to open surgery;
* Surgery planned to be performed using a single port;
* Surgery planned to be performed with a hand-assisted device;
* Requiring emergency surgery;
* Likely to require an energy tissue sealer/dissector with a shaft larger than 35cm during surgery;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants (age ≥ 18 and < 80 years of age, on the day of the procedure), scheduled to undergo a planned colectomy, anticipated to be performed laparoscopically
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of articulated activations | Intraoperative
  Number of device activations while the device is articulated

OTHER OUTCOMES:
Number and percent of perpendicular transections of vessels | Intraoperative
  Transections done at an approximate angle of 80-100 degrees, per the judgment of a third party data reviewer

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Jersey Shore University medical Center, Neptune City, New Jersey
  - The Christ Hospital, Cincinnati, Ohio

REFERENCES:
- [Result] Glenn S. Parker MD, Ben M. Tsai MD, Dipen C. Maun MD, Janice F. Rafferty MD, Michael J. Stamos MD, Edward G. Chekan MD, Michael Schwiers, and Mario Gutierrez (2015)